CLINICAL TRIAL: NCT06777758
Title: The Comparison of Remimazolam or Propofol Used Alone Versus in Combination for Moderate Sedation During Endoscopic Examination and Treatment.
Brief Title: Comparison of Remimazolam and Propofol in Endoscopic Examinations and Treatments
Acronym: Remimazolam
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Yuan-Yi Chia, Department Director, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSVGH24-CT8-16
Record Dates: First submitted 2024-12-06; First posted 2025-01-16 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Complications; Respiratory Depression; Postoperative Nausea; Vomiting; Constipation
Keywords: endoscope; Respiratory depression; Remimazolam、; Sedation; BYFAVO
MeSH Terms: conditions — Postoperative Complications; Respiratory Insufficiency; Postoperative Nausea and Vomiting; Vomiting; Constipation | interventions — remimazolam; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol (Active Comparator): The patient underwent a routine upper gastrointestinal endoscopy.
  Interventions: Drug: Propofol
- Remimazolam (Experimental): The patient underwent routine upper gastrointestinal endoscopy and Remimazolam was substituted for Propofol.
  Interventions: Drug: Remimazolam
- Propofol + Remimazolam (Experimental): The patient underwent routine upper gastrointestinal endoscopy, and the anesthetic drug used was Propofol combined with Remimazolam.
  Interventions: Drug: Remimazolam; Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam
  Arms: Propofol + Remimazolam; Remimazolam
Drug: Propofol — Propofol dose reduction ratio
  Arms: Propofol; Propofol + Remimazolam

SUMMARY:
This study aims to evaluate the efficacy and safety of Remimazolam, either used alone or in combination with Propofol, for moderate sedation anesthesia during endoscopic therapies or examinations. Additionally, it seeks to explore whether their combination can further enhance the quality of patient anesthesia and recovery outcomes.

DETAILED DESCRIPTION:
Objective This study aims to evaluate the efficacy and safety of Remimazolam, either used alone or in combination with Propofol, for moderate sedation anesthesia during endoscopic therapies or examinations. Additionally, it seeks to explore whether their combination can further enhance the quality of patient anesthesia and recovery outcomes.

Methods The investigators will conduct a prospective, randomized, single-center study. Eligible patients will be randomly allocated into three groups: the first group receiving Propofol alone for moderate sedation anesthesia (control group), the second group receiving Remimazolam alone for anesthesia, and the third group receiving a combination of Propofol and Remimazolam for anesthesia. The investigators will record anesthesia depth (DSA values of BIS), heart rate, blood pressure, oxygen saturation, and other indicators during the procedure, as well as postoperative recovery time, time to consciousness recovery, oxygen desaturation, instances of inadequate anesthesia depth, intraoperative patient movement or recall, surgeon satisfaction, patient satisfaction, readmission rate within 14 days, complications, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are between 20-80 years old.
* Anesthesiologists rated ASA as between I and III.
* Patients undergoing upper gastrointestinal endoscopic examination or therapy.

Exclusion Criteria:

* Allergy to Propofol, Remimazolam, or opioid medications.
* Emergency surgery.
* Pregnancy.
* History of malignant hyperthermia.
* Impaired liver or kidney function.
* Airway difficulties due to pharyngeal tumors.
* Refusal to participate.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose change | Perioperatively (during upper gastrointestinal endoscopy)
  Change in Propofol dose ratio. (Record total dose, Duration, mg/h/kg)

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting. | After returning to the ward from the recovery room until before breakfast on the first postoperative day.
  Track postoperative nausea and vomiting episodes.
Time to open eyes after stopping Propofol or Remimazolam. | The timer starts after the anesthetic is administered.
  Eye open minutes after Propofol or Remimazolam stop.
Use of rescue medications during surgery. | During surgery
  Rescue drugs are used during the operation
Analgesic dosage in the recovery room. | Observation period in the postoperative recovery room
  Analgesic dosage in the postoperative recovery room.
Analgesic dosage in the ward. | The patients were followed up from the time they returned to the ward after surgery to the first day after surgery.
  The dosage of analgesics used in post-operative wards.
Pain Intensity (Visual Analog Scale, VAS) every 15 minutes in the recovery room for 1 hour after surgery. | Within 1 hour post-surgery.
  Assessment of pain intensity using the Visual Analog Scale (VAS), where 0 represents no pain and 10 represents the worst possible pain.
Pain from the first injection of medication. | During the surgery (immediately after the first injection).
  Assessment of pain intensity caused by the first injection of medication, measured using the Visual Analog Scale (VAS) from 0 to 10.
Recall of surgery events. | On postoperative day 1 (within 24 hours after surgery).
  Recall events during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: CHIA-HAO YANG, M.D, Principal Investigator — employe; Tzung-Jim Tsai, M.D, Principal Investigator — employe
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Result] Meseeha M, Goosenberg E, Attia M. Endoscopic Retrograde Cholangiopancreatography. 2025 Oct 5. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK493160/ PMID 29630212
- [Result] Garewal D, Waikar P. Propofol sedation for ERCP procedures: a dilemna? Observations from an anesthesia perspective. Diagn Ther Endosc. 2012;2012:639190. doi: 10.1155/2012/639190. Epub 2012 Jan 5. PMID 22272061
- [Result] Garewal D, Vele L, Waikar P. Anaesthetic considerations for endoscopic retrograde cholangio-pancreatography procedures. Curr Opin Anaesthesiol. 2013 Aug;26(4):475-80. doi: 10.1097/ACO.0b013e3283620139. PMID 23635608
- [Result] Zhu H, Su Z, Zhou H, Lu J, Wang X, Ji Z, Chen S, Wang X, Yao M, Lu Y, Yu W, Su D. Remimazolam Dosing for Gastroscopy: A Randomized Noninferiority Trial. Anesthesiology. 2024 Mar 1;140(3):409-416. doi: 10.1097/ALN.0000000000004851. PMID 38039392
- [Result] Barbosa EC, Espirito Santo PA, Baraldo S, Meine GC. Remimazolam versus propofol for sedation in gastrointestinal endoscopic procedures: a systematic review and meta-analysis. Br J Anaesth. 2024 Jun;132(6):1219-1229. doi: 10.1016/j.bja.2024.02.005. Epub 2024 Mar 4. PMID 38443286
- [Result] Dong SA, Guo Y, Liu SS, Wu LL, Wu LN, Song K, Wang JH, Chen HR, Li WZ, Li HX, Zhang L, Yu JB. A randomized, controlled clinical trial comparing remimazolam to propofol when combined with alfentanil for sedation during ERCP procedures. J Clin Anesth. 2023 Jun;86:111077. doi: 10.1016/j.jclinane.2023.111077. Epub 2023 Feb 9. PMID 36764022
- [Result] Ahmer W, Imtiaz S, Alam DM, Ahmed K, Sajid B, Yousuf J, Asnani S, Fahim MAA, Ali R, Mansoor M, Safdar MT, Anjum MU, Hasanain M, Larik MO. Remimazolam versus propofol for sedation in gastrointestinal endoscopy and colonoscopy within elderly patients: a meta-analysis of randomized controlled trials. Eur J Clin Pharmacol. 2024 Apr;80(4):493-503. doi: 10.1007/s00228-024-03624-6. Epub 2024 Jan 23. PMID 38261005
- [Result] Rex DK, Bhandari R, Desta T, DeMicco MP, Schaeffer C, Etzkorn K, Barish CF, Pruitt R, Cash BD, Quirk D, Tiongco F, Sullivan S, Bernstein D. A phase III study evaluating the efficacy and safety of remimazolam (CNS 7056) compared with placebo and midazolam in patients undergoing colonoscopy. Gastrointest Endosc. 2018 Sep;88(3):427-437.e6. doi: 10.1016/j.gie.2018.04.2351. Epub 2018 Apr 30. PMID 29723512
- [Result] Yang SH, Wu CY, Tseng WH, Cherng WY, Hsiao TY, Cheng YJ, Chan KC. Nonintubated laryngomicrosurgery with Transnasal Humidified Rapid-Insufflation Ventilatory Exchange: A case series. J Formos Med Assoc. 2019 Jul;118(7):1138-1143. doi: 10.1016/j.jfma.2018.11.009. Epub 2018 Dec 3. PMID 30522856
- [Result] Montgomery J, Melia L, O'Donnell N, MacKenzie K. Intubation trauma and the head and neck surgeon: issues with a shared airway. J R Soc Med. 2015 Nov;108(11):426-8. doi: 10.1177/0141076815614803. No abstract available. PMID 26609095
- [Result] Kuo YT, Chang TS, Tsai CC, Chang HC, Chia YY. Optimizing nonintubated laryngeal microsurgery: The effectiveness and safety of superior laryngeal nerve block with high-flow nasal oxygen-A prospective cohort study. J Chin Med Assoc. 2024 Mar 1;87(3):334-339. doi: 10.1097/JCMA.0000000000001057. Epub 2024 Jan 30. PMID 38305707
- [Result] Lewis SR, Pritchard MW, Fawcett LJ, Punjasawadwong Y. Bispectral index for improving intraoperative awareness and early postoperative recovery in adults. Cochrane Database Syst Rev. 2019 Sep 26;9(9):CD003843. doi: 10.1002/14651858.CD003843.pub4. PMID 31557307
- [Result] Punjasawadwong Y, Phongchiewboon A, Bunchungmongkol N. Bispectral index for improving anaesthetic delivery and postoperative recovery. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD003843. doi: 10.1002/14651858.CD003843.pub3. PMID 24937564
- [Result] Wehrmann T. Extended monitoring of the sedated patient: bispectral index, Narcotrend and automated responsiveness monitor. Digestion. 2010;82(2):90-3. doi: 10.1159/000285506. Epub 2010 Apr 21. PMID 20407252
- [Result] Lee J, Jeong S, Lee DH, Park JS. Finding the ideal sedative: a non-inferiority study of remimazolam vs propofol in endoscopic retrograde cholangiopancreatography. J Gastroenterol Hepatol. 2023 Dec;38(12):2160-2166. doi: 10.1111/jgh.16354. Epub 2023 Sep 20. PMID 37730240
- [Result] Lee Y, Huang SJ, Lin PC, Lai HY, Pan MH. Low dose fentanyl and propofol improve the speed and quality of tidal-breathing induction techniques in sevoflurane anesthesia for adults. Acta Anaesthesiol Sin. 2001 Jun;39(2):83-8. PMID 11475180